CLINICAL TRIAL: NCT02401555
Title: Performance Evaluation of the Bio-Rad Geenius HIV1/2 Supplemental Assay
Status: Completed | Type: Observational
Sponsor: Bio-Rad Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: RP.BVD.GEHIV.02
Record Dates: First submitted 2015-03-16; First posted 2015-03-30 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Known HIV1 positives: Individuals known to the HIV1 positive tested with Geenius HIV1/2 Supplemental Assay
  Interventions: Device: Geenius HIV1/2 Supplemental Assay
- Known AIDS: Individuals known to meet diagnostic criteria for AIDS tested with Geenius HIV1/2 Supplemental Assay
  Interventions: Device: Geenius HIV1/2 Supplemental Assay
- Low risk (negatives): Individuals at low risk for HIV infection tested with Geenius HIV1/2 Supplemental Assay
  Interventions: Device: Geenius HIV1/2 Supplemental Assay

INTERVENTIONS:
Device: Geenius HIV1/2 Supplemental Assay — The purpose of this study is to evaluate the performance of the Bio-Rad Geenius HIV1/2 Supplemental Assay test in finger stick whole blood, venous whole blood, serum or plasma (EDTA, heparin, sodium citrate).

SUMMARY:
The purpose of this study was to evaluate the performance of the Bio-Rad Geenius HIV 1/2 Supplemental Assay, a single-use immunochromatographic assay for the confirmation and differentiation of individual antibodies to Human Immunodeficiency Virus Types 1 and 2 (HIV-1 and HIV-2) in fingerstick whole blood, venous whole blood, serum, or plasma samples (EDTA, heparin, and sodium citrate).

DETAILED DESCRIPTION:
Prospectively collected matched sample types, including fingerstick (capillary blood), serum, plasma, and whole venous blood were obtained from subjects at three clinical trial sites within the United States. Informed consent was used to enroll subjects at low risk for HIV (N=120 subjects) and from subjects pre-diagnosed as HIV positive (N=299 subjects).

The fingerstick samples were tested with Geenius HIV 1/2 Supplemental Assay at the collection site, while the remaining matched sample types, (serum, plasma, and whole venous blood) were sent to a clinical lab to be tested on the Geenius HIV 1/2 Supplemental Assay. Results of the Geenius HIV 1/2 Supplemental Assay on each of 4 matched sample were compared to the serum result on the Bio-Rad GS HIV 1/HIV 2 PLUS O EIA, Bio-Rad HIV-1 Western blot, and the Bio-Rad Multispot HIV 1/HIV-2 Rapid Test (reference methods).

Retrospective specimens from repositories or specimens purchased from commercial vendors were also included in the study. In addition to the Geenius HIV 1/2 Supplemental Assay, the GS HIV 1/HIV 2 PLUS O EIA, Bio-Rad HIV-1 Western blot, and the Bio-Rad Multispot HIV 1/HIV-2 Rapid Test were utilized as reference methods. Historical data, when available, was also used. All samples were identified with a unique study number and included the following populations/panels:

1. HIV-1/HIV-2 False Reactive Samples (N=100)
2. Unrelated Medical Conditions (N=40).
3. Normal Pediatric Patients (N=10)
4. HIV-1 Positive Pediatric Patients (N=40)
5. HIV-1 Non B Group M Subtypes (N=136)
6. HIV-1 Group O Antibody Positive (N=15)
7. Known HIV-2 Positive Population (N=200)
8. HIV Performance Panels

   1. Anti-HIV-1/2 Combo Performance Panel: PRZ208 (N=15)
   2. HIV-1 Low Titer Panel: PRB109 (N=20)
   3. HIV-1 Incidence / Prevalence Panel: PRB601 (N=15)
   4. HIV-1 Seroconversion Panels (26 Panels, N=230)
9. CEPHIA Evaluation Panel (N=2500)

ELIGIBILITY:
Inclusion Criteria for HIV1 positives and AIDS positive populations:

* Should be able to provide informed consent.
* Must be greater than or equal to 18 years of age.
* Agree to provide a finger stick sample.
* Agree to provide upto 20 mL of blood by veni-puncture.
* Must have sufficient medical history to provide data required for the case report form.

Exclusion Criteria for HIV1 positives and AIDS positive populations:

* Unable to provide informed consent
* Subjects who have received an experimental vaccine for HIV.
* Individuals except AIDS patients who are currently on ARV therapy with the duration from the start of therapy for more than 6 months.

Inclusion Criteria for Low Risk population:

* Able to provide Informed consent
* Must be greater than or equal to 18 years of age.
* Subject does not report any high risk behaviors for HIV infection.
* Of unknown HIV status.

Exclusion criteria for Low Risk Population:

* Unable to provide informed consent.
* Individuals with one or more high risk behaviors with HIV infection within the previous 6 months.
* Self reported history of HIV infection
* Prior receipt of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV1 Positives: Individuals with confirmed HIV1 positive records AIDS Positives: Individuals with proved CDC stage 3 (AIDS) Low Risk patients: Low Risk individuals including potential military recruits, soldiers and civilians who have not reported any high risk behavior for HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dennis, BS, Study Director — Bio-Rad Laboratories
Locations (5):
- United States (5):
  - HIV/AIDS Division, San Fransisco General Hospital, San Francisco, California
  - Blood Systems Research Institute, San Francisco, California
  - Center for Disease Control and Prevention, Atlanta, Georgia
  - Clinical Trials Center, Walter Reed Army Institute of Research, Silver Spring, Maryland
  - University Of Washington AIDS Clinical Trials Unit, Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Background] Delmonico FL, Snydman DR. Organ donor screening for infectious diseases: review of practice and implications for transplantation. Transplantation. 1998 Mar 15;65(5):603-10. doi: 10.1097/00007890-199803150-00001. No abstract available. PMID 9521191
- [Background] Barre-Sinoussi F, Chermann JC, Rey F, Nugeyre MT, Chamaret S, Gruest J, Dauguet C, Axler-Blin C, Vezinet-Brun F, Rouzioux C, Rozenbaum W, Montagnier L. Isolation of a T-lymphotropic retrovirus from a patient at risk for acquired immune deficiency syndrome (AIDS). Science. 1983 May 20;220(4599):868-71. doi: 10.1126/science.6189183.
- [Background] Gallo RC, Salahuddin SZ, Popovic M, Shearer GM, Kaplan M, Haynes BF, Palker TJ, Redfield R, Oleske J, Safai B, et al. Frequent detection and isolation of cytopathic retroviruses (HTLV-III) from patients with AIDS and at risk for AIDS. Science. 1984 May 4;224(4648):500-3. doi: 10.1126/science.6200936.
- [Background] Coffin J, Haase A, Levy JA, Montagnier L, Oroszlan S, Teich N, Temin H, Toyoshima K, Varmus H, Vogt P, et al. What to call the AIDS virus? Nature. 1986 May 1-7;321(6065):10. doi: 10.1038/321010a0. No abstract available. PMID 3010128
- [Background] Clavel F, Guetard D, Brun-Vezinet F, Chamaret S, Rey MA, Santos-Ferreira MO, Laurent AG, Dauguet C, Katlama C, Rouzioux C, et al. Isolation of a new human retrovirus from West African patients with AIDS. Science. 1986 Jul 18;233(4761):343-6. doi: 10.1126/science.2425430.
- [Background] Clavel F, Mansinho K, Chamaret S, Guetard D, Favier V, Nina J, Santos-Ferreira MO, Champalimaud JL, Montagnier L. Human immunodeficiency virus type 2 infection associated with AIDS in West Africa. N Engl J Med. 1987 May 7;316(19):1180-5. doi: 10.1056/NEJM198705073161903. PMID 3472076
- [Background] Centers for Disease Control (CDC). AIDS due to HIV-2 infection--New Jersey. MMWR Morb Mortal Wkly Rep. 1988 Jan 29;37(3):33-5. No abstract available. PMID 3122008
- [Background] O'Brien TR, George JR, Holmberg SD. Human immunodeficiency virus type 2 infection in the United States. Epidemiology, diagnosis, and public health implications. JAMA. 1992 May 27;267(20):2775-9. No abstract available. PMID 1578597
- [Background] Sullivan MT, Guido EA, Metler RP, Schable CA, Williams AE, Stramer SL. Identification and characterization of an HIV-2 antibody-positive blood donor in the United States. Transfusion. 1998 Feb;38(2):189-93. doi: 10.1046/j.1537-2995.1998.38298193104.x. PMID 9531953
- [Background] Brun-Vezinet F, Rey MA, Katlama C, Girard PM, Roulot D, Yeni P, Lenoble L, Clavel F, Alizon M, Gadelle S, et al. Lymphadenopathy-associated virus type 2 in AIDS and AIDS-related complex. Clinical and virological features in four patients. Lancet. 1987 Jan 17;1(8525):128-32. doi: 10.1016/s0140-6736(87)91967-2. PMID 2879971
- [Background] Quinn TC, Zacarias FR, St John RK. AIDS in the Americas: an emerging public health crises. N Engl J Med. 1989 Apr 13;320(15):1005-7. doi: 10.1056/NEJM198904133201509. No abstract available. PMID 2467206
- [Background] Guyader M, Emerman M, Sonigo P, Clavel F, Montagnier L, Alizon M. Genome organization and transactivation of the human immunodeficiency virus type 2. Nature. 1987 Apr 16-22;326(6114):662-9. doi: 10.1038/326662a0. PMID 3031510
- [Background] Janssens W, Buve A, Nkengasong JN. The puzzle of HIV-1 subtypes in Africa. AIDS. 1997 May;11(6):705-12. doi: 10.1097/00002030-199706000-00002. No abstract available. PMID 9143601
- [Background] Charneau P, Borman AM, Quillent C, Guetard D, Chamaret S, Cohen J, Remy G, Montagnier L, Clavel F. Isolation and envelope sequence of a highly divergent HIV-1 isolate: definition of a new HIV-1 group. Virology. 1994 Nov 15;205(1):247-53. doi: 10.1006/viro.1994.1640. PMID 7975221
- [Background] Simon F, Mauclere P, Roques P, Loussert-Ajaka I, Muller-Trutwin MC, Saragosti S, Georges-Courbot MC, Barre-Sinoussi F, Brun-Vezinet F. Identification of a new human immunodeficiency virus type 1 distinct from group M and group O. Nat Med. 1998 Sep;4(9):1032-7. doi: 10.1038/2017. PMID 9734396
- [Background] Meloni ST, Kim B, Sankale JL, Hamel DJ, Tovanabutra S, Mboup S, McCutchan FE, Kanki PJ. Distinct human immunodeficiency virus type 1 subtype A virus circulating in West Africa: sub-subtype A3. J Virol. 2004 Nov;78(22):12438-45. doi: 10.1128/JVI.78.22.12438-12445.2004. PMID 15507630
- [Background] Plantier JC, Leoz M, Dickerson JE, De Oliveira F, Cordonnier F, Lemee V, Damond F, Robertson DL, Simon F. A new human immunodeficiency virus derived from gorillas. Nat Med. 2009 Aug;15(8):871-2. doi: 10.1038/nm.2016. Epub 2009 Aug 2. PMID 19648927
- [Background] Gao F, Yue L, Robertson DL, Hill SC, Hui H, Biggar RJ, Neequaye AE, Whelan TM, Ho DD, Shaw GM, et al. Genetic diversity of human immunodeficiency virus type 2: evidence for distinct sequence subtypes with differences in virus biology. J Virol. 1994 Nov;68(11):7433-47. doi: 10.1128/JVI.68.11.7433-7447.1994. PMID 7933127
- [Background] George JR, Rayfield MA, Phillips S, Heyward WL, Krebs JW, Odehouri K, Soudre R, De Cock KM, Schochetman G. Efficacies of US Food and Drug Administration-licensed HIV-1-screening enzyme immunoassays for detecting antibodies to HIV-2. AIDS. 1990 Apr;4(4):321-6. doi: 10.1097/00002030-199004000-00006. PMID 2350452
- [Background] Loussert-Ajaka I, Ly TD, Chaix ML, Ingrand D, Saragosti S, Courouce AM, Brun-Vezinet F, Simon F. HIV-1/HIV-2 seronegativity in HIV-1 subtype O infected patients. Lancet. 1994 Jun 4;343(8910):1393-4. doi: 10.1016/s0140-6736(94)92524-0. PMID 7910884
- [Background] Schable C, Zekeng L, Pau CP, Hu D, Kaptue L, Gurtler L, Dondero T, Tsague JM, Schochetman G, Jaffe H, et al. Sensitivity of United States HIV antibody tests for detection of HIV-1 group O infections. Lancet. 1994 Nov 12;344(8933):1333-4. doi: 10.1016/s0140-6736(94)90695-5. PMID 7968029
- [Background] Resnick L, Veren K, Salahuddin SZ, Tondreau S, Markham PD. Stability and inactivation of HTLV-III/LAV under clinical and laboratory environments. JAMA. 1986 Apr 11;255(14):1887-91. PMID 2419594
- [Background] Bond WW, Favero MS, Petersen NJ, Ebert JW. Inactivation of hepatitis B virus by intermediate-to-high-level disinfectant chemicals. J Clin Microbiol. 1983 Sep;18(3):535-8. doi: 10.1128/jcm.18.3.535-538.1983. PMID 6630443
- [Background] Sehulster LM, Hollinger FB, Dreesman GR, Melnick JL. Immunological and biophysical alteration of hepatitis B virus antigens by sodium hypochlorite disinfection. Appl Environ Microbiol. 1981 Nov;42(5):762-7. doi: 10.1128/aem.42.5.762-767.1981. PMID 7316505
- [Background] Panlilio AL, Cardo DM, Grohskopf LA, Heneine W, Ross CS; U.S. Public Health Service. Updated U.S. Public Health Service guidelines for the management of occupational exposures to HIV and recommendations for postexposure prophylaxis. MMWR Recomm Rep. 2005 Sep 30;54(RR-9):1-17. PMID 16195697

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Known HIV1 Positives | Known AIDS | Low Risk (Negatives)
Started | 87 | 212 | 120
Completed | 87 | 212 | 120
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Known HIV1 Positives | Known AIDS | Low Risk (Negatives) | Total
Number analyzed (Participants) | 87 | 212 | 120 | 419
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 201 | 120 | 406
  >=65 years | 2 | 11 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 32 | 55 | 96
  Male | 78 | 180 | 65 | 323
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 0 | 4
  Asian | 2 | 5 | 18 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 31 | 70 | 43 | 144
  White | 45 | 119 | 56 | 220
  More than one race | 6 | 8 | 3 | 17
  Unknown or Not Reported | 2 | 4 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 87 | 212 | 120 | 419

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Result of Assay (Bio-Rad Geenius HIV 1/2 Supplemental Assay) From Accuracy Analysis
Description: The purpose of this study was to evaluate the performance of the Bio-Rad Geenius HIV1/2 Supplemental Assay, a single-use immunochromatographic assay for the confirmation and differentiation of individual antibodies to Human Immunodeficiency Virus Types1 and 2 (HIV-1 and HIV-2) in fingerstick whole blood, venous whole blood, serum, or plasma (EDTA, heparin and sodium citrate). The Accuracy analysis on the serum samples is a proportion of results that are correctly identified as such.
Time Frame: Up to 9 months
Measure: Number (95% Confidence Interval); unit: Percentage of True Results
Arm/Group | Known HIV1 Positives | Known AIDS | Low Risk (Negatives)
Number analyzed (Participants) | 87 | 212 | 120
Percentage of True Results | 100 [95.76 to 100] | 99.06 [96.62 to 99.74] | 95.83 [90.61 to 98.21]

ADVERSE EVENTS:
Time Frame: The period in which adverse event data were collected was 1 year (April 2013- April 2014).
Arm/Group | Known HIV1 Positives | Known AIDS | Low Risk (Negatives)
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/212 | 0/120
Other Adverse Events (participants affected / at risk) | 0/87 | 0/212 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a five year period from the time of the non-disclosure agreement execution.